CLINICAL TRIAL: NCT04063735
Title: Alleviating Effects Against Dry Eye by Oral Intake of Cordyceps Cicadae Mycelia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Pei-Cheng Lin (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Sponsor-Investigator, David Pei-Cheng Lin, Professor, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 16-019-A2
Record Dates: First submitted 2019-08-15; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye; Supplement
Keywords: Dry Eye; Cordyceps cicadae mycelia
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): supplement was given for 3 months.
  Interventions: Dietary Supplement: Cordyceps Cicadae Mycelia
- Placebo group (Placebo Comparator): Placebo was given for 3 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cordyceps Cicadae Mycelia — Cordyceps Cicadae Mycelia supplement for 3 months
  Arms: Experimental group
Dietary Supplement: Placebo — Placebo was given to participants.
  Arms: Placebo group

SUMMARY:
Cordyceps cicadae mycelia was tested for amelioration of dry eye symptoms through dietary supplementation. Its efficacy in relief of human dry eye status was assessed by randomized, double-blinded tests, including multiple assessments. The results were compared between the placebo group and the experimental group.

DETAILED DESCRIPTION:
Former animal studies had shown that Cordyceps cicadae mycelia can effectively ameliorate UVB-induced dry eye symptoms. This study further investigated its efficacy in human dry eye status by randomized, double-blinded tests, including dry eye questionnaires, blood tests, salivary tests, tear volume test, intra-ocular pressure assessments, ocular surface photography, corneal fluorescein stain, tear film breakup time test, fundus photography, and cornea impression cytology. All tests were performed again after 3 months of dietary supplement of either samples or placebo. A total of 97 participants completed the trial. The data were analyzed by paired-t test and compared between the placebo and the experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged from 20 to 60 with dry eye symptoms confirmed by ophthalmologists, and without chronic diseases.

Exclusion Criteria:

* Those vulnerable to damages or loss of self-conscious, or behavior capacity, or with major illness or with critical diseases.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
tear film breakup time | day 1 to day 90.
  Tear film breakup time was used for tear quality assessments.
Cornea surface scores based on Efron grading system | day 1 to day 90.
  Cornea surface scores based on Efron grading system was used for assessment of cornea surface damages.
Intra-ocular pressure | day 1 to day 90.
  Intra-ocular pressure was taken to assess eye pressure.

CONTACTS AND LOCATIONS:
Overall Officials: David Pei-Cheng Lin, PhD, Principal Investigator — Chung Shan Medical University

IPD SHARING:
Plan to Share IPD: No